CLINICAL TRIAL: NCT00933634
Title: Efficacy and Safety of Electrical Versus Pharmacological Cardioversion in Early Atrial Fibrillation: a Randomized Controlled Trial
Brief Title: Efficacy and Safety of Electrical Versus Pharmacological Cardioversion in Early Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valduce Hospital (Other)
Responsible Party: Andrea Bellone, Valduce Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECVPCV-001
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; electrical cardioversion; pharmacological cardioversion
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electric Countershock; Propafenone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- electrical cardioversion (Experimental): Patients were sedated with propofol and external cardioversion was performed in anteroposterior position (right sternal body at the third intercostal space-angle of the left scapula). Patients were submitted to a biphasic wave-form sequential shock of 100-150-200 J, if necessary.
  Interventions: Procedure: electrical cardioversion
- propafenone (Active Comparator): Propafenone (2 mg/kg bolus) was administered iv to obtain pharmacologic sinus rhythm conversion.
  Interventions: Drug: propafenone

INTERVENTIONS:
Procedure: electrical cardioversion — External cardioversion was performed in anteroposterior position (right sternal body at the third intercostal space-angle of the left scapula); patients were submitted to a biphasic wave-form sequential shock of 100-150-200 J, if necessary.
  Arms: electrical cardioversion
Drug: propafenone — Propafenone (2 mg/kg bolus) was administered to obtain pharmacolgic sinus rhythm conversion.
  Arms: propafenone

SUMMARY:
The optimal strategy to restore sinus rhythm in patients with atrial fibrillation (AF) of less than 48 hours' duration is still controversial. The investigators performed a controlled single-center trial to compare electrical and pharmacological (propafenone) cardioversion to restore the sinus rhythm in selected patients with acute atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* atrial fibrillation of less than 48 hours' duration.

Exclusion Criteria:

* AF of more than 48 hours'
* hemodynamic instability
* acute onset atrial fibrillation due to acute coronary syndrome
* electrolyte disturbances
* sepsis
* fever
* hypothermia
* untreated hyperthyroidism
* use of antiarrhythmic drugs
* high embolic risk
* unclear duration of symptoms

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of intervention (Electrical and pharmacological cardioversion) in restoring sinus rythm | during emergency department stay

SECONDARY OUTCOMES:
Number of adverse events related to electrical and pharmacological cardioversion | during emergency department stay
recurrence of atrial fibrillation | within 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Unit - Valduce Hospital, Como, Italy

REFERENCES:
- [Derived] Bellone A, Etteri M, Vettorello M, Bonetti C, Clerici D, Gini G, Maino C, Mariani M, Natalizi A, Nessi I, Rampoldi A, Colombo L. Cardioversion of acute atrial fibrillation in the emergency department: a prospective randomised trial. Emerg Med J. 2012 Mar;29(3):188-91. doi: 10.1136/emj.2010.109702. Epub 2011 Mar 21. PMID 21422032